CLINICAL TRIAL: NCT00505830
Title: Evaluation of the French Version of Screening Questionnaires for Autism and Asperger Syndrome : Autism Spectrum Quotient (AQ) Empathy Quotient (EQ) and Systemizing Quotient (SQ)
Brief Title: Evaluation of the French Version of Screening Questionnaires for Autism and Asperger Syndrome: AQ, EQ and SQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Francais d'Epidemiologie Psychiatrique (Other)
Collaborators: Joint Clinical Research Center (Other)
Other Study IDs: Autisme AQ
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Asperger Syndrome; Autism
Keywords: Asperger Syndrom; Autism Quotient; French version; screening; diagnostic test; accuracy
MeSH Terms: conditions — Asperger Syndrome; Autistic Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: 50 adolescents with AS or high functioning autism (HFS) diagnosed by psychiatrists using established criteria and with an IQ >85.
  Interventions: Other: questionnaires
- 2: 50 adolescents with AS or classical autism diagnosed by psychiatrists using established criteria 70<IQ<84.
  Interventions: Other: questionnaires
- 3: 50 adolescents with psychiatric disorders but no autism syndrom.
  Interventions: Other: questionnaires
- 4: Sample of 50 healthy adolescents selected randomly from 200.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Primary outcome:
  Autism Spectrum Quotient (AQ)
  Secondary outcome measure:
  Empathy quotient (EQ) Systemizing quotient (SQ) WISC III or WISC IV ADOS score ADI score

SUMMARY:
Autism is considered as an invading disorder of the development. Asperger Syndrome (AS) is a particular form of autism and is difficult to diagnose. The Autism Spectrum Quotient (AQ) has been developed in order to measure the degree of autistic traits in autistic adolescent with normal intelligence (Baron-Cohen et al. 2001, 2006). AQ comprises 50 questions, with 5 groups of 10 questions assessing imagination, social skills, attention switching, attention to detail and communication skills. Each of these items scores 1 point if the respondent records abnormal or autistic like behaviour. The minimum score on the AQ is 0 and the maximum 50.

The principal objective of this study is to evaluate the accuracy of the French version of Autism Spectrum Quotient questionnaire.

Secondary objectives are to:

Evaluate if EQ and SQ can distinguish adolescents without psychiatric syndromes from those with classical autism or AS.

Evaluate if AQ, EQ and SQ can distinguish adolescents with psychiatric disorders from autistic adolescents.

Define the threshold of positivity for the 3 questionnaires.

DETAILED DESCRIPTION:
4 groups of participants will be screened with the questionnaires: Group 1: 50 adolescents with AS or high functioning autism (HFS) diagnosed by psychiatrists using established criteria and with an IQ >85.

Group 2: 50 adolescents with AS or classical autism diagnosed by psychiatrists using established criteria 70<IQ<84.

Group 3: 50 adolescents with psychiatric disorders. Group 4: Sample of 50 healthy adolescents selected randomly from 200. The questionnaires are given to the parents of adolescents during the first meeting. Parents are invited to send them back to the clinical investigation centre of Lyon (France).

Multicentre study: 8 clinical centres and 18 paediatricians

ELIGIBILITY:
Inclusion Criteria:

Group 1 (AS/HFA) and 2 (AS/classic autism) :

* Boys and girls aged 12 to 18
* Patients with autism or Asperger syndrome according to the diagnostic criteria (ICD 10)
* Patients receiving education in an ordinary school
* IQ>70

Group 3 (adolescents with psychiatric disorders):

* Boys and girls aged 12 to 18
* Patients hospitalized on a psychiatric ward or at a psychiatrics patient visit or psychiatric consultation wit hout autistic syndrome
* Patients receiving education in an ordinary school when not in hospital

Group 4 (adolescent without psychiatric syndrome):

* Boys and girls aged 12 to 18
* Patients receiving education in an ordinary school

Exclusion Criteria:

For all groups :

* Problem with language or comprehension
* Participants who have not given their consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2007-07; Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Manificat, MDH, Principal Investigator — Centre Hospitalier Saint Jean de Dieu
Locations (1):
- Centre Hospitalier Saint Jean de Dieu, Lyon, France